CLINICAL TRIAL: NCT01334073
Title: Phase I Study of the Combination of Axitinib (AX) Plus Everolimus (EV) in Patients With Malignant Advanced Solid Tumors
Brief Title: Study of the Combination of Axitinib Plus Everolimus in Patients With Malignant Advanced Solid Tumors
Acronym: EVAX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/09
Record Dates: First submitted 2011-04-05; First posted 2011-04-12 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Malignant Advanced Solid Tumors; Carcinoma, Renal Cell
Keywords: Phase I; Axitinib; Everolimus; Maximum tolerated dose (MTD); solid tumor; Renal cell cancer (RCC); Pharmacokinetics (PK/PD)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib plus everolimus (Experimental)
  Interventions: Drug: Axitinib plus everolimus

INTERVENTIONS:
Drug: Axitinib plus everolimus — Patients will take both drugs orally, every day, without planned rest period (AX bid and EV once a day). By convention one cycle is 28 days. At the first cycle patients will take one week of AX single agent before starting EV. Patients will be treated at increasing dose levels (DLs) in successive cohorts of 3-6 patients according to the number of patients with dose limiting toxicities (DLT) until the maximum tolerated dose

SUMMARY:
The aim of the study is to determine the MTD of the combination of everolimus plus axitinib in solid tumors, especially RCC.

DETAILED DESCRIPTION:
Phase I study of the combination of axitinib (AX) plus everolimus (EV) in patients with malignant advanced solid tumors.

* To determine the recommended dose for phase II study of the combination of AX + EV
* To determine the safety profile and predictive factors for toxicity, pharmacokinetics (PK), and efficacy in adult solid tumors.
* To assess functional vascular imaging (FVI) as surrogate marker of activity, biomarkers predictive of activity and preliminary efficacy data in metastatic RCC, untreated with antiangiogenics.

Phase I, multicentre, open-label, non-randomized, sequential algorithm based dose-finding (3+3), clinical study in successive cohorts of patients.

Patients will take both drugs orally, every day, without planned rest period (AX bid and EV once a day). By convention one cycle is 28 days. At the first cycle patients will take one week of AX single agent before starting EV. Patients will be treated at increasing dose levels (DLs) in successive cohorts of 3-6 patients according to the number of patients with dose limiting toxicities (DLT) until the maximum tolerated dose (MTD; i.e. the DL at which <= 1/6 patient experiences a DLT during the first cycle). All decision concerning qualification for DLT, dose escalation, study termination, inclusion of additional patients, will be taken by a Trial Monitoring Committee..

The MTD will not be higher than the recommended dose of each single agent. Six additional patients will be entered at the MTD to confirm the feasibility of the dose and preliminarily assess the efficacy of the combination in patients with RCC untreated with antiangiogenics.

Three levels of dose will be explored.

ELIGIBILITY:
Inclusion criteria

* Histologically proven advanced adult solid tumors, with the exception of Hodgkin and non Hodgkin lymphoma. Patients with hepatocellular carcinomas (HCC) may be enrolled without histological documentation if they meet the consensus non-invasive diagnostic criteria.
* Failure or contra-indication of all standard therapies, except for the patients with advanced renal cell carcinoma, enrolled at the recommended dose who will be naïve of previous lines of therapy while metastatic.
* Age > 18 years
* ECOG Performance status (PS) 0-1
* Life expectancy > 3 months
* Measurable/evaluable disease according to RECIST CRITERIA version 1.0
* Acceptable biological values: Hemoglobin > 10g /dL; neutrophils > 1.5 x 109/L; platelets > 100 x 109/L, AST and ALT < 2.5 x the upper normal limits (UNL), or < 5 x UNL in case of liver metastases, GGT < 3 x the upper normal limits (UNL), PAL < 2.5 x the upper normal limits (UNL), or < 5 x UNL in case of liver metastases, serum bilirubin < 1.5 x ULN, creatinine clearance (Cockroft & Gault formula) > 60 mL/min.
* 24 hours proteinuria ≤ 1 g/24 h
* Albumin > 30 g/l
* Amylase and lipase ≤ 1.5 UNL
* Electrolytes (calcium, sodium, potassium, chlore, magnesium, phosphate) in the normal range. Supplementation could be possible before study entry.
* Total cholesterol ≤ 2.5 UNL
* Triglycerides ≤ 2.5 UNL
* BP < 140/90
* Washout period from last anticancer therapy, including radiation and surgery > 3 weeks and recovery of toxicities to NCI-CTC grade < 1.
* Written informed Consent.
* Use of effective contraceptive method (Intrauterine device, oral combined contraceptive) for women of child-bearing age or whose partner is included in the trial.
* Patient with french social security.
* Additional inclusion criteria before the association axitinib plus everolimus period
* No toxicity with NCI-CTC grade > 2 at the end of axitinib alone period just before starting axitinib and everolimus (cycle 1)
* BP < 140/ 90

Exclusion criteria

* Brain metastasis
* Severe underlying cardiovascular disease, even medically controlled, such as angina pectoris, myocardial infarction, cardiac insufficiency, cardiac failure, cerebral strokes, lower limb ischemic disease, thromboembolic disease, and any patient, who, in the investigator's opinion is at high risk for arterial or venous thromboembolism.
* Hepatitis B or C carrier or at a chronic state
* Uncontrolled hypertension, or diabetes mellitus despite medical treatment.
* Inability to swallow pills
* Unresolved pneumopathy, no need for antibiotherapy
* Any medical or social condition, which; in the investigator's opinion, would jeopardize patient's safety, patient's compliance to the protocol, or the interpretation of study results. These conditions include (but are not limited to): severe infection, cardiac failure, chronic gastrointestinal disease compromising oral drug absorption, psychiatric illnesses, foreseeable poor treatment compliance with oral medications, patients living far away from the investigational centers, etc…
* Hypersensitivity to Axitinib or Everolimus
* Participation to another clinical trial, or use of an unapproved medication within 4 weeks prior to study treatment initiation.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with DLT (dose limiting toxicity) during the first cycle (first 28 days of the combination of both study compounds), per dose level explored | during cycle 1
  A DLT will be one of the following adverse events, with a possible relationship to the study medications
  * Febrile, related bleeding or any grade 4 neutropenia or thrombocytopenia,
  * grade 3 non-hematological toxicity, unless adequately treated with usual symptomatic therapy
  * grade 4 non-hematological toxicity
  * study treatment interruption > 2 weeks, inability to deliver at least 80% of the intended doses of axitinib and/or everolimus between day 8 and 35 due to toxicity.

SECONDARY OUTCOMES:
Adverse event (AE) will be graded according to NCI-CTC criteria V3 | After each cycle of treatement
  Number of AE per patient, per grade, per cycle and per dose level, proportion
Best response rate will be assessed according to RECIST criteria, during the follow-up | Every other cycle of treatment
  Frequency (total, per dose level), proportion
Rate of non-tumor progression at 16 weeks | at 16 weeks
  Frequency (total, per dose level), proportion
Progression-free Survival (PFS) defined as the time between study treatment initiation and either tumor progression or death, regardless of the cause, whichever occurs first and PFS at 1 year | 1 year
  Frequency (total, per dose level), probability
Comparison of PK parameters | day 1 (axitinib alone) and day 15 (everolimus combined with axitinib)
  Plasma PK using peak concentration (Cmax), area under the concentration versus time curve (AUC), volume of distribution at steady state (Vdss), plasma clearance (CL) and plasma half-life (t1/2). PK parameters will be compared to severe (grade 3-4) AEs, tumor responses and non-tumor progression at 16 weeks. PK parameters of axitinib combined to everolimus (day 15) will be compared to PK parameters of axitinib alone in the same patient (day 1). PK of everolimus combined to axitinib (day 15) will be compared to historical data of everolimus alone

CONTACTS AND LOCATIONS:
Overall Officials: Alain RAVAUD, Principal Investigator — University Hospital, Bordeaux; Adélaïde Doussau, Dr, Study Chair — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Professeur Alain RAVAUD, Bordeaux
  - Professeur Jean-Pierre DELORD, Toulouse

REFERENCES:
- [Background] Su Y, Amiri KI, Horton LW, Yu Y, Ayers GD, Koehler E, Kelley MC, Puzanov I, Richmond A, Sosman JA. A phase I trial of bortezomib with temozolomide in patients with advanced melanoma: toxicities, antitumor effects, and modulation of therapeutic targets. Clin Cancer Res. 2010 Jan 1;16(1):348-57. doi: 10.1158/1078-0432.CCR-09-2087. Epub 2009 Dec 22. PMID 20028756
- [Background] O'Reilly T, Lane HA, Wood JM, Schnell C, Littlewood-Evans A, Brueggen J, McSheehy PM. Everolimus and PTK/ZK show synergistic growth inhibition in the orthotopic BL16/BL6 murine melanoma model. Cancer Chemother Pharmacol. 2011 Jan;67(1):193-200. doi: 10.1007/s00280-010-1307-z. Epub 2010 May 30. PMID 20512579
- [Background] Choueiri TK. Axitinib, a novel anti-angiogenic drug with promising activity in various solid tumors. Curr Opin Investig Drugs. 2008 Jun;9(6):658-71. PMID 18516765